CLINICAL TRIAL: NCT03287401
Title: Prediction of Postoperative Anesthesia Care Unit Delirium Using Electroencephalography - German Validation Study
Brief Title: Prediction of PACU Delirium Using EEG - German Validation Study
Acronym: PACUD-EEG
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: PACUD-EEG
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Delirium
Keywords: EEG; PACU Delirium
MeSH Terms: conditions — Delirium | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with general anesthesia: Patients with general anaesthesia are monitored with electroencephalography and the results will be associated with the risk for PACU delirium
  Interventions: Device: Electroencephalography

INTERVENTIONS:
Device: Electroencephalography — Patients electroencephalogram will be recorded

SUMMARY:
Aim of this observational study is to investigate whether frontal electroencephalogram analysis is able to predict increased risk for PACU delirium.

DETAILED DESCRIPTION:
Delirium in the postoperative anaesthesia care unit (PACU), a special of form of postoperative delirium, is associated with increased hospital stay and an elevated hospital re-admission rate. First studies investigating the patients' electroencephalogram (EEG) on emergence from anaesthesia were able to show that an abrupt change of predominant EEG-rhythm is associated with an increased rate of PACU delirium. Therefore, it seems possible to use frontal EEG in order to identify patients being at elevated risk for PACU delirium.

Aim of this observational study is to validate the results of an international collaboration in a German population of patients undergoing general anaesthesia. EEG in these patients is recorded from start of anaesthesia until emergence. Rate of PACU delirium is assessed using the CAM-ICU score 15 and 60 minutes after emergence in the recovery room.

In a pilot study in 626 patients from 2013 to 2015 in 5 international study centres the rate of PACU delirium was 20%. As it is planned to investigate 5 co-factors using regression analysis 50 cases of delirium will be necessary for a sufficient analysis. Therefore, in total 250 patients will be included.

Due to an additional study centre that included 50 patients enrolment of the german validation group was completed after 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 years or older
* surgery in general anaesthesia

Exclusion Criteria:

* emergency surgery
* general anaesthesia within 30 days before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients above the age of 18 years undergoing general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
PACU Delirium | Emergence from anaesthesia until discharge from postoperative anaesthesia care unit (60 minutes)
  Detection of delirium in the postoperative anaesthesia care unit using CAM-ICU score

SECONDARY OUTCOMES:
Pain in the PACU (NRS) | Emergence from anaesthesia until discharge from postoperative anaesthesia care unit (60 minutes)
  Pain assessed with numeric rating scale
Electroencephalography | Pre-induction until emergence from anaesthesia (average of 3 hours)
  Electroencephalography recording

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Schmid, MD, Principal Investigator — Klinikum rechts der Isar - Dept. of Anaesthesiology
Locations (1):
- Klinikum rechts der Isar Dept. of Anesthesiology, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Derived] Lutz R, Muller C, Dragovic S, Schneider F, Ribbe K, Anders M, Schmid S, Garcia PS, Schneider G, Kreuzer M, Kratzer S. The absence of dominant alpha-oscillatory EEG activity during emergence from delta-dominant anesthesia predicts neurocognitive impairment- results from a prospective observational trial. J Clin Anesth. 2022 Nov;82:110949. doi: 10.1016/j.jclinane.2022.110949. Epub 2022 Aug 29. PMID 36049381